CLINICAL TRIAL: NCT02575014
Title: Preoperative Hyperbaric Oxygen Therapy (HBOT) vs. Non Preoperative HBOT in Patients Undergoing Pancreaticoduodenectomy for Premalignant, and Malignant Tumors of the Common Bile Duct, Periampullary and Duodenum
Brief Title: Pancreaticoduodenectomy With or Without Preoperative Hyperbaric Oxygen Therapy
Acronym: HBOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Florida Hospital Tampa Bay Division (Other)
Responsible Party: Principal Investigator, Alexander Rosemurgy, Director, Surgical Digestive Disorders and GERD Center, Director HPB Surgery and Fellowship Program, Florida Hospital Tampa Bay Division
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HBOT 529762
Record Dates: First submitted 2015-10-07; First posted 2015-10-14 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Periampullary Tumor; Common Bile Duct Neoplasms; Duodenal Neoplasms
MeSH Terms: conditions — Common Bile Duct Neoplasms; Duodenal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperative HBOT (Experimental): 25 out of 50 patients will receive 2 preoperative hyperbaric oxygen therapy treatments, one the day before their operation, the other within 5 hours preceding their operation. The participants will be treated with up to 2.4 ATA O2, for a maximum of 90 minutes each day with or without air breaks, as deemed necessary by the investigator. Day 0 will be the first day of their HBOT treatment, Day 1 will be the day of their operation and second/final HBOT treatment.
  Interventions: Drug: Preoperative hyperbaric oxygen
- No HBOT (No Intervention): 25 out of 50 patients will not receive preoperative hyperbaric oxygen therapy. Day 1 will be the day of the operation.

INTERVENTIONS:
Drug: Preoperative hyperbaric oxygen — Subjects undergoing preoperative HBOT will be treated with up to 2.4 ATA O2, for a maximum of 90 minutes each day with or without air breaks, as deemed necessary by the investigator, for two days. The two days will be the day of and the day immediately prior to the operation.
  Other Names: O2
  Arms: Preoperative HBOT

SUMMARY:
The primary objective of this study is to assess the safety, tolerability and toxicity of preoperative HBOT in patients undergoing a pancreaticoduodenal resection for premalignant and malignant tumors of the common bile duct, periampullary and duodenum.

DETAILED DESCRIPTION:
Patients diagnosed with premalignant and malignant tumors of the common bile duct, periampullary and duodenum will be screened for eligibility within 4 weeks of their scheduled surgery. Initiation of therapy is defined as the first day of HBOT for patients receiving HBOT therapy (Arm A) and the day of surgery for patients not receiving HBOT (Arm B). Patients will be considered "enrolled into study" once the consent form has been signed, all screening procedures have been undertaken and all the eligibility criteria are met. The fifty eligible patients will be randomized in a 1:1 ratio the same day of the screening process. The eligible subjects undergoing HBOT will be treated with up to 2.4 Atmospheres Absolute (ATA) of oxygen (O2), for a maximum of 90 minutes each day with or without air breaks, as deemed necessary by the investigator, for two days. Patients who are deemed ineligible will receive the same standard of care without any exceptions. The start day of the week to commence HBOT will be Monday through Wednesday, as the second and final day of HBOT treatment will be the day in which the patient undergoes pancreaticoduodenectomy. The subjects who complete the HBOT regimen must undergo subsequent pancreaticoduodenectomy within five hours of termination of HBOT. If there is more than a five hour delay from completion of the HBOT to commencement of operation, the subject will be considered "off study treatment". However, "off study treatment" patients will continue to be followed up every six months for the first thirty months, and annually thereafter. During the postoperative period, clinical data and questionnaire forms will be collected on day 1, day 3, day 5, and one month (± 2 weeks) during the first year. As for secondary objectives, the investigators will collect clinical data from patients during their follow up visits in the office, by contacting them on the phone, or by mailing them the protocol specific questionnaires every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed via endoscopic ultrasound (EUS) and fine needle aspiration (FNA) or CT-guided biopsy with periampullary adenocarcinoma, duodenal cancer, premalignant lesions of the pancreas (pancreatic intraepithelial neoplasia, intraductal papillary mucinous neoplasm) and cholangiocarcinoma (Klatskin tumor) undergoing pancreaticoduodenectomy
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2
* One or more comorbidities:

Diabetes Mellitus Chronic Obstructive Pulmonary Disease Cardiac Disease: history of angina, myocardial infarction, previous percutaneous cardiac intervention, or cardiac surgery, dysrhythmia Peripheral Vascular Disease: history of revascularization or amputation, rest pain, or gangrene Neurological Disease: history of stroke with or without residual deficit, seizure disorder, transient ischemic attack, hemiplegia, paraplegia, or impaired sensorium Dyspnea Bleeding Disorder Metabolic Disease (e.g. BMI ≥ 35) Renal Insufficiency Hepatic Insufficiency Another comorbidity that in the opinion of the investigator makes the patient compromised

* Nutritionally depleted. Albumin level ≤ 3.5 grams/deciliter (g/dL)
* Adequate organ function defined as:

Absolute neutrophil count >1,500 / (microliter) mcL Platelets >100,000 / mcL Total bilirubin <2.5 time upper limits of normal Aspartate aminotransferase (AST) / Alanine transaminase (ALT) <2.5 times institutional upper limit of normal Creatinine within normal institutional limits OR creatinine clearance >60 mL/min/ per Cockcroft-Gault equation for patients with creatinine levels above institutional normal

- Signed informed consent

Exclusion Criteria:

* History of asthma. There is some evidence that the administration of some bronchodilators may increase the incidence of gas embolism to the brain through pulmonary vasodilation.
* Congenital spherocytosis. Increased risk of massive hemolysis.
* High grade fever at time of screening (more than 38.5 degree Celsius tend to lower the seizure threshold due to oxygen toxicity and may result in the delay of relatively routine therapy
* Optic neuritis.
* Upper respiratory tract infection and viral infection (relative contra-indications due to the difficulty such patients may have in clearing their ears and sinuses.
* Pregnancy.
* Emphysema with carbon dioxide retention.
* Viral infection. There are controversial clinical evidences whether the hyperbaric oxygen therapy (HBOT) can be helpful in eliminating viral infections or otherwise viral infections may be considerably worsened after HBOT.
* Cisplatin therapy (some evidence that this drug retards wound healing when combined with HBOT).
* Disulphiram therapy. Evidence suggests that this drug blocks the production of superoxide dismutase. This may severely affect the body's ability to neutralize oxygen free radicals.
* Doxorubicin therapy. This chemotherapeutic agent becomes increasingly toxic under pressure. Animal studies suggest at least a one-week break between last dose and first treatment of HBOT.
* Claustrophobia. Some degree of confinement anxiety has been reported.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with hyperbaric oxygen treatment related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Preoperative
  ear pain, oxygen toxicity, visual changes, embolism, pneumothorax, fatigue

SECONDARY OUTCOMES:
Death | Postoperative up to 5 years
Length of hospital stay | Postoperative up to one month
Postoperative complications | Postoperative up to one month
  Surgical wound infections, hernia, abscess, fluid collection, bleeding, anastomotic leak, thromboembolic events, pulmonary atelectasis, bronchospasm, pneumonia, stroke, myocardial ischemia, myocardial infarction, time to extubation for patients requiring prolonged mechanical assistance, biliary or pancreatic fistula, fever, blood transfusion, delayed gastric emptying,
Change in Interleukin-2 | Postoperative up to one month
Change in Interleukin-6 | Postoperative up to one month
Change in Interleukin-10 | Postoperative up to one month
Change in Vascular Endothelial Growth Factor | Postoperative up to one month
Change in Transforming Growth Factor-Beta | Postoperative up to one month
Change in Erythrocyte Sedimentation Rate | Postoperative up to one month
Change in Quality of Life QOL-C30 v1.0 | Postoperative up to 5 years
  Postoperative quality of life scores will be compared to preoperative quality of life
Change in pain score according to visual analog scale | Postoperative up to one month
  Postoperative pain will be compared to preoperative pain
Change in Cancer Antigen 19-9 | Postoperative up to one year
Change in Carcinoembryonic antigen | Postoperative up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Rosemurgy, MD, Principal Investigator — Florida Hospital Tampa
Locations (1):
- Florida Hospital Tampa, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No